CLINICAL TRIAL: NCT01106846
Title: Analgesic Effect of Ketamine in Patients Undergoing Hysteroscopic Endometrial Thermal Ablation Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Resources not available to complete.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Shireen Ahmad, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STU00026695
Record Dates: First submitted 2010-04-16; First posted 2010-04-20 (Estimated); Results first posted 2015-07-20 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-07

CONDITIONS: Pain
Keywords: Ketamine; Anesthesia; Pain; Outpatient surgery
MeSH Terms: conditions — Pain | interventions — Sodium Chloride; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: Saline group (Placebo Comparator): Group A: Saline group , infusion of saline intravenously
  Interventions: Drug: Group A: Saline Group
- Group B: 1% Ketamine group (Active Comparator): Group B: Infusion of ketamine 1% intravenously
  Interventions: Drug: Group B: 1% Ketamine group

INTERVENTIONS:
Drug: Group A: Saline Group — Saline continuous infusion
  Other Names: Saline
  Arms: Group A: Saline group
Drug: Group B: 1% Ketamine group — Administration of 1% ketamine intravenously.
  Other Names: Ketamine
  Arms: Group B: 1% Ketamine group

SUMMARY:
Hypothesis: The intraoperative administration of ketamine will result in a 30% reduction in opiate requirement following endometrial ablation surgery and the intraoperative administration of ketamine will result in a decreased time to meet discharge criteria in the PACU following endometrial ablation surgery.

The research question is "Does intraoperative administration of ketamine result in decreased postoperative opiate requirement and time to discharge from the postanesthesia recovery unit (PACU) following hysteroscopic endometrial ablation".

DETAILED DESCRIPTION:
Preoperatively:

Subjects will be recruited up to 21days prior to the day of surgery. After informed consent is obtained, subjects will be randomly assigned to one of two groups:

Group A: Saline group Group B: 1% Ketamine group

A verbal rating scale (VRS) will be used to assess pain preoperatively. The patient will be asked to identify the severity of pain by indicating on a scale of 0-10 where 0 is "no pain" and 10 is "the worst pain imaginable".

Baseline Quality of Recovery will be obtained. (Appendix F)

Subjects will be randomized prior to surgery to either Group A or Group B. The randomization table is computer generated. There is a 50% allocation to each group.

Intraoperatively:

Standard anesthetic monitoring will be used including monitoring of processed EEG including either the bi-spectral index (BIS) or similar standard of care ASA monitor. A standardized intraoperative anesthetic plan will be utilized by the anesthesia personnel. (Appendix A). Study drug will be prepared and labeled in 10mL syringes by research personnel who will not be involved in the study assessments. Study drug will be administered on initial insertion of Novasure® device (Appendix B).

Postoperatively:

Pain scores in the PACU will be assessed using the VRS upon admission and every 30 minutes thereafter until discharge criteria are met.

Additionally, nausea, vomiting and retching episodes will be recorded using a VRS.

Postoperative analgesic and antiemetic therapy will be standardized and total amounts of these agents will be recorded Assessment of psychomimetic effects including sedation and agitation will be assess postoperatively prior to discharge using the Richmond Agitation/Sedation Scale (Appendix D).

Acute recovery will be assessed using the Modified Post Anesthesia Discharge Scoring System (MPADSS) (Appendix E). A score of 8 or greater will indicate discharge readiness. Time to fulfill discharge criteria will be recorded.

Any other adverse events and medications required will be recorded. These data will be recorded by research personnel who will be blinded to the study group assignments.

Subjects will be contacted by telephone 24 hours after surgery to assess post-discharge quality of recovery (Appendix F).

ELIGIBILITY:
Inclusion Criteria:

* Gender: Female
* Age: 18-65 years
* Non-pregnant, non-lactating
* Surgery: Outpatient hysteroscopic Novasure® endometrial ablation
* Language: English speaking
* Consent: Obtained

Exclusion Criteria:

* Patient refusal
* Under 18 or over age 65
* Non-English Speaking
* Pregnancy, Breast feeding
* Hysteroscopic procedures using Thermachoice® ablation device
* Chronic use or addiction to opiates, sedatives, non-opiate analgesics
* History of heavy alcohol usage (>4 drinks/day)
* Significant cardiovascular or pulmonary disease
* Psychiatric or emotional disorder
* Allergy to anesthetic agents utilized in the protocol
* Glaucoma
* Thyrotoxicosis

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shireen Ahmad, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Prentice Women's Hosptial, Chicago, Illinois

REFERENCES:
- [Background] Schenker JG, Margalioth EJ. Intrauterine adhesions: an updated appraisal. Fertil Steril. 1982 May;37(5):593-610. doi: 10.1016/s0015-0282(16)46268-0. No abstract available. PMID 6281085
- [Background] Jansen FW, Vredevoogd CB, van Ulzen K, Hermans J, Trimbos JB, Trimbos-Kemper TC. Complications of hysteroscopy: a prospective, multicenter study. Obstet Gynecol. 2000 Aug;96(2):266-70. doi: 10.1016/s0029-7844(00)00865-6. PMID 10908775
- [Background] Wong AY, Wong K, Tang LC. Stepwise pain score analysis of the effect of local lignocaine on outpatient hysteroscopy: a randomized, double-blind, placebo-controlled trial. Fertil Steril. 2000 Jun;73(6):1234-7. doi: 10.1016/s0015-0282(00)00498-2. PMID 10856489
- [Background] Lau WC, Ho RY, Tsang MK, Yuen PM. Patient's acceptance of outpatient hysteroscopy. Gynecol Obstet Invest. 1999;47(3):191-3. doi: 10.1159/000010092. PMID 10087415
- [Background] De Iaco P, Marabini A, Stefanetti M, Del Vecchio C, Bovicelli L. Acceptability and pain of outpatient hysteroscopy. J Am Assoc Gynecol Laparosc. 2000 Feb;7(1):71-5. doi: 10.1016/s1074-3804(00)80012-2. PMID 10648742
- [Background] MacPherson RD, Woods D, Penfold J. Ketamine and midazolam delivered by patient-controlled analgesia in relieving pain associated with burns dressings. Clin J Pain. 2008 Sep;24(7):568-71. doi: 10.1097/AJP.0b013e31816cdb20. PMID 18716494
- [Background] White PF, Way WL, Trevor AJ. Ketamine--its pharmacology and therapeutic uses. Anesthesiology. 1982 Feb;56(2):119-36. doi: 10.1097/00000542-198202000-00007. No abstract available. PMID 6892475
- [Background] Bowdle TA, Radant AD, Cowley DS, Kharasch ED, Strassman RJ, Roy-Byrne PP. Psychedelic effects of ketamine in healthy volunteers: relationship to steady-state plasma concentrations. Anesthesiology. 1998 Jan;88(1):82-8. doi: 10.1097/00000542-199801000-00015. PMID 9447860
- [Background] Deng XM, Xiao WJ, Luo MP, Tang GZ, Xu KL. The use of midazolam and small-dose ketamine for sedation and analgesia during local anesthesia. Anesth Analg. 2001 Nov;93(5):1174-7. doi: 10.1097/00000539-200111000-00023. PMID 11682390

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of recruitment 03/15/2010-02/14/2013.
Period: Overall Study
Arm/Group | Group A: Saline Group | Group B: 1% Ketamine Group
Started | 12 | 10
Completed | 12 | 9
Not Completed | 0 | 1
Not completed — Change in surgical procedure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Saline Group | Group B: 1% Ketamine Group | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 22
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.08 (3.88) | 43.12 (6.19) | 44.28 (4.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Quality of Recovery Score Post Operative at 24 Hours
Description: Quality of recovery 40 score at 24 hours after the surgical procedure. 40 being a poor recovery and 200 being a good recovery.
Time Frame: 24 hours post operative
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Group A: Saline Group | Group B: 1% Ketamine Group
Number analyzed (Participants) | 12 | 9
units on scale | 191.2 (9.15) | 191.1 (11.3)
Statistical Analysis 1: Comparison: Group A: Saline Group vs Group B: 1% Ketamine Group; Test type: Superiority or Other; p = .947, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 Hour post operative
Arm/Group | Group A: Saline Group | Group B: 1% Ketamine Group
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 3/12 | 0/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Saline Group (N=12) | Group B: 1% Ketamine Group (N=9)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) — Nausea 60 minutes post operative

LIMITATIONS AND CAVEATS:
Study was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes